CLINICAL TRIAL: NCT02750046
Title: Collection of Bone Specimens for Testing of A Special Vessel Subtype
Brief Title: Study of A Special Vessel Subtype in Bone Samples From Patients With Osteoporotic and Nonosteoporotic Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SencondSoochowU
Record Dates: First submitted 2016-03-24; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- osteoporotic fractures (Experimental): patients with osteoporotic fractures, including femoral neck fracture and pertrochanteric fracture. Total hip arthroplasty or proximal femoral nails was needed.
  Interventions: Procedure: total hip arthroplasty or proximal femoral nails
- nonosteoporotic fractures (Sham Comparator): patients with nonosteoporotic fractures, including femoral neck fracture and pertrochanteric fracture. Total hip arthroplasty or proximal femoral nails was needed.
  Interventions: Procedure: total hip arthroplasty or proximal femoral nails

INTERVENTIONS:
Procedure: total hip arthroplasty or proximal femoral nails — Bone samples from Hip fracture were collected when total hip arthroplasty or proximal femoral nails was performed.

SUMMARY:
RATIONALE: Collecting and storing bone samples from patients with osteoporotic and nonosteoporotic fracture to study a special vessel subtype in the laboratory may help surgeon learn more about the relationship between bone mineral density (BMD) and a special vessel subtype (type H vessel).

PURPOSE: This research study is looking at changes of a special vessel subtype in bone samples from patients with osteoporotic and nonosteoporotic fracture.

DETAILED DESCRIPTION:
OBJECTIVES:

1. Establish type H vessel in bone specimen in patients with hip fracture.
2. Explore the correlation of BMD and type H vessel.

OUTLINE:

1. Collect human bone specimens from patients with Osteoporotic and Nonosteoporotic Fracture.
2. Provide a repository for storage of tissue and make these specimens available for approved projects by laboratory-based investigators.
3. Observe the type H vessel in bone slice by immunofluorescence staining.
4. Collect clinical data on these patients including bone mineral density.
5. Investigate the relationship between BMD and type H vessel.

ELIGIBILITY:
Inclusion Criteria:

1. Ages Eligible for Study: 65-75 Years
2. Genders Eligible for Study: Woman
3. Accepts Healthy Volunteers: NO
4. Study Population: Female patients with hip fracture. -

Exclusion Criteria:

1. Malignancy or benign ovarian cysts
2. Known chronic or systemic diseases
3. Hormone therapy in the previous 3 months
4. Bone metabolism and drug therapy

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
The area of a special vessel subtype in human bone samples | 3 months
  Bone samples were fixed in 4% PFA, decalcified, dehydrated, embedded and immunofluorescent staining for 3 months. Calculate the proportion of the special vessel of total vessel.

SECONDARY OUTCOMES:
The value of bone mineral density | 1 week
  Bone mineral density was measured by double energy X-ray absorptiometer (DXA) in a week before surgery.
Correlation of of bone mineral density and area of a special vessel subtype in human bone | 2 months
  Calculate correlation coefficient of BMD and type H vessel in human bone samples in 2 months.

CONTACTS AND LOCATIONS:
Overall Officials: Youjia Xu, PhD. M.D., Study Chair — Second Affiliated Hospital of Soochow University
Locations (1):
- Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kusumbe AP, Ramasamy SK, Adams RH. Coupling of angiogenesis and osteogenesis by a specific vessel subtype in bone. Nature. 2014 Mar 20;507(7492):323-328. doi: 10.1038/nature13145. Epub 2014 Mar 12. PMID 24646994
- [Result] Xie H, Cui Z, Wang L, Xia Z, Hu Y, Xian L, Li C, Xie L, Crane J, Wan M, Zhen G, Bian Q, Yu B, Chang W, Qiu T, Pickarski M, Duong LT, Windle JJ, Luo X, Liao E, Cao X. PDGF-BB secreted by preosteoclasts induces angiogenesis during coupling with osteogenesis. Nat Med. 2014 Nov;20(11):1270-8. doi: 10.1038/nm.3668. Epub 2014 Oct 5. PMID 25282358
- [Result] Ramasamy SK, Kusumbe AP, Wang L, Adams RH. Endothelial Notch activity promotes angiogenesis and osteogenesis in bone. Nature. 2014 Mar 20;507(7492):376-380. doi: 10.1038/nature13146. Epub 2014 Mar 12. PMID 24647000
- [Result] Kusumbe AP, Adams RH. Osteoclast progenitors promote bone vascularization and osteogenesis. Nat Med. 2014 Nov;20(11):1238-40. doi: 10.1038/nm.3747. No abstract available. PMID 25375923
- [Derived] Wang L, Zhou F, Zhang P, Wang H, Qu Z, Jia P, Yao Z, Shen G, Li G, Zhao G, Li J, Mao Y, Xie Z, Xu W, Xu Y, Xu Y. Human type H vessels are a sensitive biomarker of bone mass. Cell Death Dis. 2017 May 4;8(5):e2760. doi: 10.1038/cddis.2017.36. PMID 28471445